CLINICAL TRIAL: NCT04633187
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Effects of EDP-938 in Hematopoietic Cell Transplant Recipients With Acute Respiratory Syncytial Virus Infection of the Upper Respiratory Tract
Brief Title: Effects of EDP-938 in Hematopoietic Cell Transplant Recipients Infected With Respiratory Syncytial Virus of the Upper Respiratory Tract
Acronym: RSVTx
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to a strategic business decision and not due to safety concerns.
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDP 938-103
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-07

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — EDP-938

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EDP-938 (Experimental)
  Interventions: Drug: EDP-938
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-938 — EDP-938 800mg
  Dose adjustments were made for subjects taking azole antifungals.
  Arms: EDP-938
Drug: Placebo — Subjects took EDP-938 matching placebo tablets once a day orally for 21 days
  Arms: Placebo

SUMMARY:
This was a Phase 2b, randomized, double-blind, placebo-controlled, multicenter study evaluating the efficacy and safety of EDP-938 in HCT recipients with acute RSV infection and symptoms of URTI.

ELIGIBILITY:
Inclusion Criteria:

* Received an autologous HCT (within 6 months of signing ICF) or an allogeneic HCT (any time) using any conditioning regimen
* Absolute lymphocyte count (ALC) <500 cells/ µL in allogeneic HCT recipients. Absolute lymphocyte count (ALC) <300 cells/ µL in autologous HCT recipients.
* Laboratory confirmed RSV diagnosis from a respiratory sample obtained within 3 days before signing the ICF.
* New onset of at least one of the following respiratory symptoms within 3 days before signing the ICF: nasopharyngeal discharge, nasopharyngeal congestion, sneezing, sinus congestion, sore throat, hoarseness, earache, cough, shortness of breath, respiratory wheeze, or worsening of one of these symptoms if present chronically (associated with a previously existing diagnosis [eg, chronic rhinorrhea, chronic lung disease]) in the 3 days before signing the ICF or at Screening.
* No evidence of new abnormalities consistent with LRTI on a chest imaging (chest x-ray and/or computed tomography) performed in the 2 days before signing the ICF or at the Screening visit if there is no chest X-ray and/or computed tomography available in the 2 days before signing the ICF.
* Oxygen saturation >95% on room air.
* A woman of childbearing potential who is sexually active with a male must agree to use two effective methods of contraception from the date of Screening until 30 days after her last dose of study drug.
* A male subject who has not had a vasectomy and is sexually active with a woman of childbearing potential must agree to use effective contraception from the date of Screening to 90 days after his last dose of study drug.

Exclusion Criteria:

* Admitted to the hospital primarily for a lower respiratory tract disease of any cause as determined by the Investigator.
* Known to be concurrently infected with other respiratory viruses (eg, severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2] or other coronavirus, influenza, parainfluenza, human rhinovirus, adenovirus, human metapneumovirus) within 7 days before signing the ICF, as determined by local testing.
* Clinically significant viremia, bacteremia, or fungemia, or bacterial or fungal pneumonia within 2 weeks before signing the ICF that has not been adequately treated, as determined by the Investigator.
* Known positive human immunodeficiency virus (HIV).
* Any clinical manifestation resulting in QT prolongation.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (64):
- Augusta University Medical Center, Augusta, Georgia, United States
- Argentina (4):
  - Fundación Favaloro, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Instituto Fides, La Plata, Ciudad Autónoma de BuenosAires
  - Sanatorio Allende S.A., Córdoba, Córdoba Province
  - Hospital Britanico de Buenos Aires, Buenos Aires
- Belgium (3):
  - UZ Antwerpen, Edegem, Antwerpen
  - Institute Jules Bordet, Anderlecht, Brussels Capital
  - Hôpital de Jolimont, La Louvière
- Brazil (6):
  - Chronos Pesquisa Clínica, Brasília, Federal District
  - Hospital de Clinicas de Porto Alegre (HCPA) - PPDS, Porto Alegre, Rio Grande do Sul
  - Hospital Universitário de Santa Maria, Santa Maria, Rio Grande do Sul
  - Fundação PIO XII, Barretos, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
- Toronto General Hospital, Toronto, Ontario, Canada
- Queen Mary Hospital, Hong Kong, Hong Kong, China
- Hospital Pablo Tobón Uribe, Medellín, Colombia
- France (5):
  - CHU de Nice, Nice, Alpes-Maritimes
  - Hôtel Dieu -Angers, Angers, Maine-et-Loire
  - Hôpital Claude Huriez, Lille, Nord
  - Hopital Cote de Nacre, Caen
  - Hôpital Saint Antoine, Paris
- Greece (2):
  - Attikon University General Hospital, Athens
  - Evangelismos General Hospital of Athens, Athens
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (6):
  - ASST degli Spedali Civili di Brescia - Spedali Civili di Brescia - INCIPIT - PIN, Brescia, Lombardy
  - A.O.U. Maggiore della Carità, Novara, Piedmont
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona-Umberto I G.M. Lancisi G. Salesi, Ancona, The Marches
  - Azienda ULSS 8 "Berica" - Ospedale San Bortolo, Vicenza, Veneto
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione Policlinico Universitario A Gemelli, Roma
- Instituto Nacional de Cancerologia, Mexico City, Mexico
- Poland (2):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy Oddzial w Gliwi, Gliwice, Silesian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk
- South Africa (3):
  - Albert Alberts Stem Cell Transplant Centre, Pretoria, Gauteng
  - FCRN Clinical Trial Centre (Pty) Ldt, Vereeniging, Gauteng
  - WITS Clinical Research Site, Johannesburg
- South Korea (5):
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Gachon University Gil Medical Center, Ulsan
- Spain (13):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital de San Pedro de Alcantara, Cáceres, Caceres
  - Hospital Universitario Virgen de La Arrixaca, El Palmar, Murcia
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Regional Universitario de Malaga - Hospital General, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (2):
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Changhua
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (3):
  - Ege Universitesi Tip Fakultesi Hastanesi, Bornova, İzmir
  - Namik Kemal University, Tekirdağ, Tekirdağ
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
- Imperial College, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- EDP-938: EDP-938 150mg/400mg/800mg
- Placebo: Placebo
Period: Overall Study
Arm/Group | EDP-938 | Placebo
Started | 5 | 4
EDP-938 150 mg | 1 | 0
EDP-938 400 mg | 1 | 0
EDP-938 800 mg | 3 | 0
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- EDP-938: EDP-938: EDP-938 150/400/800mg
  The EDP-938 doses were adjusted to account for inhibitory effects of Azole antifungals on hepatic metabolism, and EDP-938 doses of 150mg and 400mg; when EDP-938 is co-administered with azole antifungals that are strong or moderate CYP3A4 inhibitors, respectively, provide similar exposures to the 800mg dose
- Total: Total of all reporting groups
Arm/Group | EDP-938 | Placebo | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.4 (15.98) | 44.3 (15.99) | 44.3 (14.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Develop Lower Respiratory Tract (LRTC) Complication
Time Frame: Day 1 through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | EDP-938 | Placebo
Number analyzed (Participants) | 5 | 4
Participants | 0 | 1

2. Secondary Outcome: Change From Baseline in RSV RNA Viral Load
Time Frame: Day 1 through Day 49
Population: Six participants (3 in each treatment group) had detectable RSV by RT-qPCR at baseline and were included in the mITT by RT-qPCR analysis population.
Measure: Mean (Standard Deviation); unit: RSV viral load (log10 copies/mL)
Arm/Group | EDP-938 | Placebo
Number analyzed (Participants) | 3 | 3
RSV viral load (log10 copies/mL) | -7.072 (0.7738) | -2.221 (6.8552)

3. Secondary Outcome: Proportion of Subjects Progressing to Respiratory Failure (of Any Cause) Requiring Mechanical Ventilation (Invasive or Noninvasive) or All-cause Mortality
Time Frame: Day 1 through Day 49
Measure: Count of Participants; unit: Participants
Arm/Group | EDP-938 | Placebo
Number analyzed (Participants) | 5 | 4
Participants | 0 | 0

4. Secondary Outcome: Safety as Measured the Number of Participants With at Least One Treatment-emergent Adverse Event
Time Frame: Day 1 through Day 49
Measure: Count of Participants; unit: Participants
Arm/Group | EDP-938 | Placebo
Number analyzed (Participants) | 5 | 4
Participants | 5 | 3

5. Secondary Outcome: Plasma PK Concentrations of EDP-938 800mg
Time Frame: Day 1 Predose and Postdose, Day 4 Predose, Day 7 Predose and Postdose, Day 11 Predose, Day 16 Predose, Day 21 Predose and Postdose
Population: Pharmacokinetic (PK) Population, PK data for subjects who received EDP-938 800 mg doses. If more than 50% of subjects have post dose concentration values below the limit of quantification (BLQ), descriptive statistics are not presented.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- EDP-938: EDP-938: EDP-938 800mg
  The EDP-938 doses were adjusted to account for inhibitory effects of Azole antifungals on hepatic metabolism, and EDP-938 doses of 150mg and 400mg; when EDP-938 is co-administered with azole antifungals that are strong or moderate CYP3A4 inhibitors, respectively, provide similar exposures to the 800mg dose.
Arm/Group | EDP-938
Number analyzed (Participants) | 3
ng/mL
  Day 1 Predose | 0 (0)
  Day 1 Postdose | 1123.33 (1028.899)
  Day 4 Predose | 1610.00 (175.784)
  Day 7 Predose | 1342.33 (411.554)
  Day 7 Postdose | 1394.33 (493.504)
  Day 11 Predose | 1176.67 (204.287)
  Day 16 Predose | 860.00 (411.887)
  Day 21 Predose | 755.33 (58.011)
  Day 21 Postdose | 1136.00 (656.195)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected beginning on Day 1 and concluded at the End-of-Study (EOS) visit on Day 49, 28 days following the last dose of the study drug.
Description: The EDP-938 doses were adjusted to account for inhibitory effects of Azole antifungals on hepatic metabolism, and EDP-938 doses of 150mg and 400mg; when EDP-938 is co-administered with azole antifungals that are strong or moderate CYP3A4 inhibitors, respectively, provide similar exposures to the 800mg dose. Adverse Events are presented for all dosages combined because, as noted above, subjects had an equivalent exposure across all EDP-938 doses administered.
Arm/Group | EDP-938 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 4/5 | 0/4
Other Adverse Events (participants affected / at risk) | 5/5 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EDP-938 (N=5) | Placebo (N=4)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EDP-938 (N=5) | Placebo (N=4)
Cellulitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Cytomegalovirus hepatitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 0
Epstein-Barr virus infection reactivation (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Calcium deficiency (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Vitamin C deficiency (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Zinc deficiency (Metabolism and nutrition disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0
Intensive care unit acquired weakness (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigators and the Sponsor that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT04633187/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT04633187/SAP_001.pdf